CLINICAL TRIAL: NCT02532855
Title: A Phase III, Multicenter, Randomized, Double-Blind, Active-Comparator Controlled Clinical Trial to Study the Safety and Efficacy of the Addition of Sitagliptin Compared With the Addition of Dapagliflozin in Subjects With Type 2 Diabetes Mellitus and Mild Renal Impairment Who Have Inadequate Glycemic Control on Metformin With or Without a Sulfonylurea
Brief Title: A Study to Assess the Addition of Sitagliptin to Metformin Compared With the Addition of Dapagliflozin to Metformin in Participants With Type 2 Diabetes Mellitus (T2DM) and Mild Renal Impairment Who Have Inadequate Glycemic Control on Metformin With or Without a Sulfonylurea (MK-0431-838)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0431-838; 2014-005525-13 (EudraCT Number); MK-0431-838 (Other: Merck Protocol Number)
Record Dates: First submitted 2015-08-25; First posted 2015-08-26 (Estimated); Results first posted 2018-10-10 (Actual); Last update posted 2018-11-20 (Actual); Status verified 2018-10

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate; dapagliflozin; Metformin; Sulfonylurea Compounds

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sitagliptin (Experimental): Participants receive sitagliptin 100 mg once daily plus matching placebo for dapagliflozin 5 mg once daily for 4 weeks followed by sitagliptin 100 mg once daily plus matching placebo for dapagliflozin 10 mg once daily for 20 weeks. Participants continue pre-study metformin (at least 1500 mg daily) alone or in combination with a sulfonylurea agent (at a dose of ≥ 50% maximum labeled dose in the country of the investigational site) throughout the duration of the study.
  Interventions: Drug: Sitagliptin; Drug: Metformin; Drug: Matching placebo to dapagliflozin; Drug: Sulfonylurea
- Dapagliflozin (Active Comparator): Participants receive dapagliflozin 5 mg once daily plus matching placebo for sitagliptin 100 mg once daily for 4 weeks followed by dapagliflozin 10 mg once daily plus matching placebo for sitagliptin 100 mg once daily for 20 weeks. Participants continue pre-study metformin (at least 1500 mg daily) alone or in combination with a sulfonylurea agent (at a dose of ≥ 50% maximum labeled dose in the country of the investigational site) throughout the duration of the study.
  Interventions: Drug: Dapagliflozin; Drug: Metformin; Drug: Matching placebo to sitagliptin; Drug: Sulfonylurea

INTERVENTIONS:
Drug: Sitagliptin — Sitagliptin 100 mg oral tablet
  Arms: Sitagliptin
Drug: Dapagliflozin — Dapagliflozin 5 mg or 10 mg oral capsule. Up-titration to dapagliflozin 10 mg daily may be delayed if participant is unable to tolerate up-titration in the opinion of the investigator. Dapagliflozin 10 mg daily may be down-titrated to dapagliflozin 5 mg daily if participant is unable to tolerate the higher dose in the opinion of the investigator.
  Arms: Dapagliflozin
Drug: Metformin — This medication is a standard-of-care medication and is administered in an open-label fashion. Supply of background metformin oral tablet(s) (at least 1500 mg daily) will be the responsibility of the participant throughout the duration of the study.
Drug: Matching placebo to sitagliptin — Matching placebo to sitagliptin 100 mg oral tablet
  Arms: Dapagliflozin
Drug: Matching placebo to dapagliflozin — Matching placebo to dapagliflozin 5 mg or 10 mg oral capsule. Up-titration to matching placebo to dapagliflozin 10 mg daily may be delayed if participant is unable to tolerate up-titration in the opinion of the investigator. Matching placebo to dapagliflozin 10 mg daily may be down-titrated to matching placebo to dapagliflozin 5 mg daily if participant is unable to tolerate the higher dose in the opinion of the investigator.
  Arms: Sitagliptin
Drug: Sulfonylurea — This medication is a standard-of-care medication and is administered in an open-label fashion. The dose of the sulfonylurea agent will be required to be at least 50% of maximum labeled dose, consistent with near maximum efficacy of the sulfonylurea agent.

SUMMARY:
The purpose of the study is to assess the effect of the addition of sitagliptin to metformin with or without a sulfonylurea compared with the addition of dapagliflozin to metformin with or without a sulfonylurea on hemoglobin A1c (A1C) over 24 weeks of treatment as well as the overall safety and tolerability of sitagliptin in comparison to that of dapagliflozin after 24 weeks of treatment. The primary hypothesis is that the change from baseline in A1C in participants treated with the addition of sitagliptin is non-inferior compared to that in participants treated with the addition of dapagliflozin after 24 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria

* Have T2DM at Screening visit
* Be on metformin monotherapy ≥1500 mg/day alone or in combination with an sulfonylurea agent (at a dose of ≥ 50% maximum labeled dose in the country of the investigational site) for ≥8 weeks
* Is a male or a female not of reproductive potential (defined as one who is postmenopausal or has had a hysterectomy and/or bilateral oophorectomy, or had bilateral tubal ligation or occlusion at least 6 weeks prior to Screening visit). If participant is a female of reproductive potential, must agree to remain abstinent from heterosexual activity or agrees to use (or have her partner use) acceptable contraception to prevent pregnancy while receiving blinded study drug and for 14 days after the last dose of blinded study drug

Exclusion Criteria:

* Has a history of type 1 diabetes mellitus or a history of ketoacidosis
* Has a history of secondary causes of diabetes
* Has a known hypersensitivity or intolerance to any dipeptidyl peptidase IV (DPP-4) inhibitor or sodium-glucose cotransporter 2 (SGLT2) inhibitor
* Has been treated with any anti-hyperglycemic agents (AHA) other than metformin and for participants on dual combination therapy, a sulfonylurea within 12 weeks of screening
* Intends to initiate weight loss medication during the study period
* Has undergone bariatric surgery within 12 months of Screening visit
* Has started a weight loss medication or a medication associated with weight changes within the prior 12 weeks.
* Has a history of myocardial infarction, unstable angina, arterial revascularization, stroke, transient ischemic attack, heart failure within 3 months of Screening visit
* Has a history of malignancy ≤5 years prior to study, except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer
* Has human immunodeficiency virus (HIV)
* Has blood dyscrasias or any disorders causing hemolysis or unstable red blood cells, or clinically important hematological disorder (such as aplastic anemia, myeloproliferative or myelodysplastic syndromes, thrombocytopenia)
* Has a medical history of active liver disease (other than non-alcoholic hepatic steatosis), including chronic hepatitis B or C, primary biliary cirrhosis, or symptomatic gallbladder disease
* Is currently being treated for hyperthyroidism or is on thyroid replacement therapy and has not been on a stable dose for at least 6 weeks prior to Screening visit
* Is on or likely to require treatment for ≥14 consecutive days or repeated courses of corticosteroids
* Is on or likely to require treatment for ≥7 consecutive days with non-steroidal anti-inflammatory drugs
* Is pregnant or breast-feeding, or is planning to conceive during the study, including 14 days following the last dose of blinded study drug
* Is planning to undergo hormonal therapy in preparation to donate eggs during the study, including 14 days following the last dose of blinded study drug
* Routinely consumes >2 alcoholic drinks per day or >14 alcoholic drinks per week or engages in binge drinking
* Has donated blood or blood products within 6 weeks of Screening visit or who plans to donate blood or blood products at any time during the study

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 614 (Actual)
Dates: Start 2015-10-20 (Actual); Primary Completion 2017-10-10 (Actual); Study Completion 2017-10-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Natale P, Tunnicliffe DJ, Toyama T, Palmer SC, Saglimbene VM, Ruospo M, Gargano L, Stallone G, Gesualdo L, Strippoli GF. Sodium-glucose co-transporter protein 2 (SGLT2) inhibitors for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2024 May 21;5(5):CD015588. doi: 10.1002/14651858.CD015588.pub2. PMID 38770818
- [Derived] Scott R, Morgan J, Zimmer Z, Lam RLH, O'Neill EA, Kaufman KD, Engel SS, Raji A. A randomized clinical trial of the efficacy and safety of sitagliptin compared with dapagliflozin in patients with type 2 diabetes mellitus and mild renal insufficiency: The CompoSIT-R study. Diabetes Obes Metab. 2018 Dec;20(12):2876-2884. doi: 10.1111/dom.13473. Epub 2018 Aug 16. PMID 30019498

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 183 medical centers in 24 countries.
Pre-assignment Details: Male and female participants, 25 years or older, with Type 2 diabetes mellitus (T2DM) and mild renal impairment on metformin alone or in combination with a sulfonylurea (SU) agent were enrolled in this trial.
Period: Overall Study
Arm/Group | Sitagliptin | Dapagliflozin
Started | 307 | 307
Treated | 307 | 306 (One participant had a protocol violation, was randomized but did not take study medication.)
Completed | 299 | 296
Not Completed | 8 | 11
Not completed — Lost to Follow-up | 4 | 3
Not completed — Withdrawal by Subject | 4 | 8

BASELINE CHARACTERISTICS:
Population: All randomized and treated participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Sitagliptin | Dapagliflozin | Total
Number analyzed (Participants) | 307 | 306 | 613
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: All randomized and treated participants
  Years | 67.7 (8.5) | 66.6 (8.6) | 67.1 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: All randomized and treated participants
  Participants
    Female | 138 | 120 | 258
    Male | 169 | 186 | 355
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: All randomized and treated participants
  Participants
    American Indian or Alaska Native | 18 | 14 | 32
    Asian | 11 | 7 | 18
    Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
    Black or African American | 8 | 11 | 19
    White | 240 | 234 | 474
    More than one race | 30 | 39 | 69
    Unknown or Not Reported | 0 | 0 | 0
Hemoglobin A1C [Mean (Standard Deviation); unit: Percent A1C] — Population: All randomized and treated participants
  Percent A1C | 7.7 (0.7) | 7.8 (0.7) | 7.7 (0.7)
Fasting Plasma Glucose (FPG) [Mean (Standard Deviation); unit: mg/dL] — Population: All randomized and treated participants
  mg/dL | 162.3 (40.4) | 165.2 (40.6) | 163.8 (40.5)
Background Antihyperglycemic Agent (AHA) [Count of Participants; unit: Participants] — Population: All randomized and treated participants
  Participants
    Metformin Alone | 212 | 225 | 437
    Metformin and Sulfonylurea | 95 | 81 | 176
Incremental 2-hour Postprandial Glucose Excursion (PPGE) [Mean (Standard Deviation); unit: mg/dL] — The PPGE is the increment (mean increase) in glucose from T-0 (T=0 minutes) to T-120 (T=120 minutes) after eating the standard meal. The PPGE was analyzed for participants who underwent the 2-point or 3-point Mixed Meal Tolerance Test (MMTT). Blood samples were drawn immediately prior to (T-0) and 60 (T-60) and 120 minutes (T-120) after a standard meal. Population: All randomized and treated participants who underwent MMTT analysis and had a baseline measurement for this endpoint.
  mg/dL
    number analyzed (Participants) | 295 | 290 | 585
    (all) | 96.2 (55.3) | 95.7 (47.1) | 95.9 (51.4)
2-hr Postprandial Glucose [Mean (Standard Deviation); unit: mg/dL] — The 2-hour postprandial glucose was analyzed for participants who underwent the 2-point or 3-point MMTT. Blood samples were drawn immediately prior to (T-0) and 60 (T-60) and 120 minutes (T-120) after a standard meal. Population: All randomized and treated participants who underwent MMTT analysis and had a baseline measurement for this endpoint.
  mg/dL
    number analyzed (Participants) | 296 | 292 | 588
    (all) | 257.7 (67.1) | 259.9 (64.4) | 258.8 (65.7)
Glucagon Area Under the Curve (AUC0-120 minutes) [Mean (Standard Deviation); unit: pmol.hr/L] — The glucagon area under the curve AUC endpoints were analyzed for participants who underwent the 3-point MMTT. Blood samples were drawn immediately prior to (T-0) and 60 (T-60) and 120 minutes (T-120) after a standard meal. The AUC curve was generated with the 3 time points. Population: All randomized and treated participants who underwent MMTT analysis and had a baseline measurement for this endpoint.
  pmol.hr/L
    number analyzed (Participants) | 108 | 109 | 217
    (all) | 49.6 (44.7) | 51.8 (45.1) | 50.7 (44.8)
Insulin AUC0-120 minutes [Mean (Standard Deviation); unit: mIU.hr/L] — The insulin area under the curve AUC endpoints were analyzed for participants who underwent the 3-point MMTT. Blood samples were drawn immediately prior to (T-0) and 60 (T-60) and 120 minutes (T-120) after a standard meal. The AUC curve was generated with the 3 time points. Population: All randomized and treated participants who underwent MMTT analysis and had a baseline measurement for this endpoint.
  mIU.hr/L
    number analyzed (Participants) | 113 | 112 | 225
    (all) | 155.0 (121.8) | 139.9 (93.5) | 147.5 (108.7)
Insulin AUC0-120 minutes to Glucagon AUC0-120 minutes Ratio [Mean (Standard Deviation); unit: Ratio] — The insulin to glucagon AUC ratio endpoint was analyzed for participants who underwent the 3-point MMTT. Blood samples were drawn immediately prior to (T-0) and 60 (T-60) and 120 minutes (T-120) after a standard meal. The AUC curve was generated with the 3 time points Population: All randomized and treated participants who underwent MMTT analysis and had a baseline measurement for this endpoint.
  Ratio
    number analyzed (Participants) | 104 | 102 | 206
    (all) | 4.0 (3.7) | 3.5 (3.0) | 3.8 (3.4)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in A1C at Week 24
Description: A1C is blood marker used to report average blood glucose levels over prolonged periods of time. Percentage A1C is the ratio of glycated hemoglobin to total hemoglobin x 100. Thus, this change from baseline reflects the Week 24 A1C minus the Week 0 A1C.
Time Frame: Baseline and Week 24
Population: All randomized and treated participants who had at least one observation for the analysis endpoint, at baseline or subsequent to at least one dose of study treatment.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent A1C
Arm/Group | Sitagliptin | Dapagliflozin
Number analyzed (Participants) | 307 | 306
Percent A1C | -0.51 [-0.60 to -0.43] | -0.36 [-0.45 to -0.27]
Statistical Analysis 1: Comparison: Sitagliptin vs Dapagliflozin; Test type: Non-Inferiority — For the primary hypothesis, sitagliptin will be considered non-inferior to dapagliflozin if the upper bound of the two-sided 95% confidence interval (CI) of the between-group difference in least squares mean change from baseline in A1C (sitagliptin minus dapagliflozin) is less than 0.3% (the non-inferiority margin). Longitudinal data analysis (LDA), Antihyperglycemic agent (AHA), Least squares means (LSM); LDA model including terms for treatment, time, background AHA, the interaction of time and background AHA, and the interaction of time by treatment; Difference in LSM (Sit. - Dap.) = -0.15, 95% CI 2-sided [-0.26 to -0.04]
Statistical Analysis 2: Comparison: Sitagliptin vs Dapagliflozin; Test type: Superiority; p = 0.006, Longitudinal data analysis; [statistical method as in outcome 1, analysis 1]; Difference in LSM (Sit. - Dap.) = -0.15, 95% CI 2-sided [-0.26 to -0.04]

2. Primary Outcome: Percentage of Participants Who Experienced One or More Adverse Events
Description: An adverse event (AE) is any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product. The AE does not have to have a causal relationship with this treatment. The AE can include any unfavourable and unintended sign, symptom, or disease or any worsening (change in frequency and/or intensity) of a preexisting condition that is temporally associated with the use of the pharmaceutical product.
Time Frame: Up to 26 weeks
Population: All randomized and treated participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Sitagliptin | Dapagliflozin
Number analyzed (Participants) | 307 | 306
Percentage of participants | 48.9 | 51.6
Statistical Analysis 1: Comparison: Sitagliptin vs Dapagliflozin; Test type: Other; Miettinen & Nurminen method; Difference in % (Sit. - Dap.) = -2.8, 95% CI 2-sided [-10.7 to 5.1]

3. Primary Outcome: Percentage of Participants Who Discontinued Study Drug Due to an AE
Description: as for outcome 2
Time Frame: Up to 24 weeks
Population: All randomized and treated participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Sitagliptin | Dapagliflozin
Number analyzed (Participants) | 307 | 306
Percentage of participants | 3.3 | 3.3
Statistical Analysis 1: Comparison: Sitagliptin vs Dapagliflozin; Test type: Other; Miettinen & Nurminen method; Difference in % (Sit. - Dap.) = -0.0, 95% CI 2-sided [-3.0 to 3.0]

4. Secondary Outcome: Change From Baseline in Incremental 2-hour (2-hr) Postprandial Glucose Excursion (PPGE) at Week 24
Description: The 2hr PPGE is the change from baseline in the mean incremental change in post meal glucose defined as T-120 minus T-0 for each participant: change from baseline PPGE = Week 24 mean (T-120 minus T-0) minus Baseline mean (T-120 minus T-0). The 2-point MMTT measured values at T-0 and T-120 while the 3-point MMTT measured values at T-0, T-60, and T-120: although only a subset of the study had the 3-point MMTT performed, all participants had a T-0 and T-120 time point. A negative (-) change from baseline to Week 24 indicates better control of postprandial glucose.
Time Frame: Immediately before and 120 minutes after the standard meal at Baseline and Week 24
Population: All randomized and treated participants who underwent MMTT for the analysis endpoint, had both baseline and Week 24 endpoint measurements, without: drug compliance <75%, use of prohibited AHA medications or pharmacologic doses of corticosteroids or incorrect double-blind study drug or a change in metformin or sulfonylurea dose.
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Sitagliptin | Dapagliflozin
Number analyzed (Participants) | 298 | 296
mg/dL | -24.2 [-30.4 to -18.0] | -18.5 [-24.9 to -12.1]
Statistical Analysis 1: Comparison: Sitagliptin vs Dapagliflozin; Test type: Superiority; p = 0.138, LDA; [statistical method as in outcome 1, analysis 1]; Difference in LSM (Sit. - Dap.) = -5.7, 95% CI 2-sided [-13.3 to 1.8]

5. Secondary Outcome: Change From Baseline in 2-hr Postprandial Glucose (PPG) at Week 24
Description: The 2hr PPG is the change from baseline in mean post prandial glucose (change from baseline PPG = Week 24 mean T-120 glucose minus Baseline mean T-120 glucose) and shows each drugs impact on PPG. The 2-point MMTT measured values at T-0 and T-120 while the 3-point MMTT measured values at T-0, T-60, and T-120: although only a subset of the study had the 3-point MMTT performed, all participants had a T-0 and T-120 time point. A negative (-) change from baseline to Week 24 indicates better control of postprandial glucose.
Time Frame: Immediately before and 120 minutes after the standard meal at Baseline and Week 24
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Sitagliptin | Dapagliflozin
Number analyzed (Participants) | 258 | 248
mg/dL | -40.4 [-46.9 to -33.9] | -37.0 [-43.7 to -30.3]
Statistical Analysis 1: Comparison: Sitagliptin vs Dapagliflozin; Test type: Superiority; The ANCOVA model included terms for treatment, background AHA, and the baseline 2-hour PPG value as a covariate; Difference in the LSM (Sit. - Dap.) = -3.4, 95% CI 2-sided [-12.1 to 5.3]

6. Secondary Outcome: Change From Baseline in Glucagon Area Under the Curve (AUC0-120 Minutes) at Week 24
Description: AUC endpoints were analyzed for participants who underwent the 3-point MMTT. Blood samples were drawn immediately prior to (T=0 minutes) and 60 and 120 minutes after the administration of the standard meal. The AUC curve was generated with the 3 time points. If any time point for a given participant was missing, the AUC was not included. Change in Postprandial Glucagon AUC after the morning meal (t=0 to 120 minutes) was calculated from the glucagon AUC over the first 120 minutes following the morning meal at baseline minus glucagon AUC over the first 120 minutes following the morning meal at Week 24. A negative (-) change from baseline to Week 24 indicates better control of postprandial glucose.
Time Frame: Immediately before and 60 and 120 minutes after the standard meal at Baseline and Week 24
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: pmol.hr/L
Arm/Group | Sitagliptin | Dapagliflozin
Number analyzed (Participants) | 85 | 88
pmol.hr/L | -4.2 [-8.8 to 0.4] | 0.2 [-4.4 to 4.8]
Statistical Analysis 1: Comparison: Sitagliptin vs Dapagliflozin; Test type: Superiority; The ANCOVA model included terms for treatment, background AHA, and the baseline glucagon AUC value as a covariate; Difference in the LSM (Sit. - Dap.) = -4.4, 95% CI 2-sided [-10.1 to 1.4]

7. Secondary Outcome: Change From Baseline in Insulin AUC0-120 Minutes at Week 24
Description: AUC endpoints were analyzed for participants who underwent the 3-point MMTT. Blood samples were drawn immediately prior to (T=0 minutes) and 60 and 120 minutes after the administration of the standard meal. The AUC curve was generated with the 3 time points. If any time point for a given participant was missing, the AUC was not included. Change in Postprandial Insulin AUC after the morning meal (t=0 to 120 minutes) was calculated from insulin AUC over the first 120 minutes following the morning meal at baseline minus insulin AUC over the first 120 minutes following the morning meal at Week 24. A negative (-) change from baseline to Week 24 indicates better control of postprandial glucose.
Time Frame: Immediately before and 60 and 120 minutes after the standard meal at Baseline and Week 24
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: mIU.hr/L
Arm/Group | Sitagliptin | Dapagliflozin
Number analyzed (Participants) | 96 | 94
mIU.hr/L | -23.4 [-36.8 to -9.9] | -28.2 [-42.1 to -14.4]
Statistical Analysis 1: Comparison: Sitagliptin vs Dapagliflozin; Test type: Superiority; The ANCOVA model included terms for treatment, background AHA, and the baseline insulin AUC value as a covariate; Difference in the LSM (Sit. - Dap.) = 4.9, 95% CI 2-sided [-12.2 to 22.0]

8. Secondary Outcome: Change From Baseline in Postprandial Insulin AUC0-120 Minutes to Glucagon AUC0-120 Minutes Ratio at Week 24
Description: AUC endpoints were analyzed for participants who underwent the 3-point MMTT. Blood samples were drawn immediately prior to (T=0 minutes) and 60 and 120 minutes after the administration of the standard meal. The AUC curve was generated with the 3 time points. If any time point for a given participant was missing, the AUC was not included. The endpoint was calculated from the ratio of (insulin AUC / glucagon AUC) over the first 120 minutes following the morning meal at baseline minus AUC over the first 120 minutes following the morning meal at Week 24. A negative (-) change from baseline to Week 24 indicates better control of postprandial glucose.
Time Frame: Immediately before and 60 and 120 minutes after the standard meal at Baseline and Week 24
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Sitagliptin | Dapagliflozin
Number analyzed (Participants) | 83 | 81
Ratio | -0.6 [-1.1 to -0.0] | -1.2 [-1.8 to -0.7]
Statistical Analysis 1: Comparison: Sitagliptin vs Dapagliflozin; Test type: Superiority; The ANCOVA model included terms for treatment, background AHA, and the baseline insulin AUC to glucagon AUC ratio value as a covariate; Difference in the LSM (Sit. - Dap.) = 0.6, 95% CI 2-sided [-0.1 to 1.3]

9. Secondary Outcome: Percentage of Participants With A1C <7% (53 mmol/Mol) at Week 24
Description: A1C is blood marker used to report average blood glucose levels over prolonged periods of time and is reported as a percentage (%). Percentage A1C is the ratio of glycated hemoglobin to total hemoglobin x 100.
Time Frame: Week 24
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Sitagliptin | Dapagliflozin
Number analyzed (Participants) | 307 | 306
Percentage of Participants | 42.6 | 27.0
Statistical Analysis 1: Comparison: Sitagliptin vs Dapagliflozin; Test type: Other — The percentage of participants was estimated using standard multiple imputation techniques from LDA model including terms for treatment, time, background AHA, the interaction of time and background AHA, and the interaction of time by treatment; Miettinen and Nurminen (M&N) method with multiple imputation from a LDA Model; Difference in % (Sit. - Dap.) = 15.5, 95% CI 2-sided [7.7 to 23.2]

10. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 24
Description: Blood glucose was measured on a fasting basis. Blood was drawn at predose on Day 1 and after 24 weeks of treatment to determine change in plasma glucose levels (i.e., FPG at Week 24 minus FPG at Week 0).
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Sitagliptin | Dapagliflozin
Number analyzed (Participants) | 307 | 306
mg/dL | -16.5 [-20.6 to -12.5] | -20.1 [-24.3 to -15.9]
Statistical Analysis 1: Comparison: Sitagliptin vs Dapagliflozin; Test type: Superiority; [statistical method as in outcome 1, analysis 1]; Difference in the LSM (Sit. - Dap.) = 3.5, 95% CI 2-sided [-1.2 to 8.3]

ADVERSE EVENTS:
Time Frame: Up to 26 weeks
Description: An AE is any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not have to have a causal relationship. The AE can include any unfavourable and unintended sign, symptom, or disease or any worsening (change in frequency and/or intensity) of a preexisting condition that is temporally associated with the use of the pharmaceutical product. The population analyzed included all randomized and treated participants.
Arm/Group | Sitagliptin | Dapagliflozin
All-Cause Mortality (participants affected / at risk) | 0/307 | 0/306
Serious Adverse Events (participants affected / at risk) | 10/307 | 13/306
Other Adverse Events (participants affected / at risk) | 22/307 | 21/306
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sitagliptin (N=307) | Dapagliflozin (N=306)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Sinus node dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1)
Reflux gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Atypical pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Epiphyseal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Partial seizures (Nervous system disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sitagliptin (N=307) | Dapagliflozin (N=306)
Hypoglycaemia (Metabolism and nutrition disorders) | 22 (51) | 21 (64)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-15): https://cdn.clinicaltrials.gov/large-docs/55/NCT02532855/Prot_SAP_000.pdf